CLINICAL TRIAL: NCT06223230
Title: Nutritional Psychological Intervention and Vomit-free Management on Survival and Quality of Life in Advanced Gastrointestinal Tumors
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Renmin Hospital of Wuhan University (Other)
Responsible Party: Principal Investigator, Yongshun Chen, Professor, Renmin Hospital of Wuhan University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: WDRY2022-K092
Record Dates: First submitted 2024-01-16; First posted 2024-01-25 (Actual); Last update posted 2024-01-30 (Actual); Status verified 2024-01

CONDITIONS: Digestive System Cancer; Digestive System Neoplasm
MeSH Terms: conditions — Digestive System Neoplasms

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study group (Experimental): First-line treatment received standard antitumor therapy and nutritional psychological interventions with and without vomit management
  Interventions: Other: Nutritional psychological interventions and vomit-free management
- Control group (No Intervention): First-line treatment receives standard antitumor therapy

INTERVENTIONS:
Other: Nutritional psychological interventions and vomit-free management — Nutritional psychological interventions and vomit-free management
  Arms: Study group

SUMMARY:
Aims to observe and evaluate the impact of survival and quality of life of patients with gastrointestinal tumors such as advanced esophageal, gastric, liver, pancreatic, and colorectal cancers through nutritional-psychological interventions versus no-vomit management compared to standard antitumor therapy alone

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-75, male or female;
2. Patients with advanced esophageal cancer, gastric cancer, liver cancer and colorectal cancer and other gastrointestinal tumors diagnosed by pathological histology or cytology;
3. Expected survival ³ 8 weeks and able to receive long-term follow-up;
4. Eastern Cooperative Oncology Group(ECOG)-Performance Status(PS) score of 0-2;
5. First-line treatment receiving standard oncology treatment and nutritional psychological intervention and vomit-free management group (study group); first-line treatment receiving only standard oncology treatment group (control group);
6. Voluntarily signing an informed consent form.

Exclusion Criteria:

1. Other malignant tumors diagnosed within the previous 5 years, except for effectively treated basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or effectively resected in situ cervical cancer or breast cancer;
2. history of psychiatric illness prior to the diagnosis of the tumor
3. patients who resist treatment
4. patients with poorly controlled severe heart disease, liver or kidney insufficiency, severe anemia, multiple lymph node enlargement, leukopenia, etc;
5. patients who are pregnant or have a pregnancy plan;
6. patients who, in the judgment of the investigator, are not suitable for inclusion in this study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 316 (Estimated)
Dates: Start 2022-06-01 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Median progression-free survival time | Approximately 40 months from date of the first participant randomization
  Progression-free survival is defined as the period from the date of treatment to the date of the first occurrence of disease progression or death from any cause, whichever occurs first. Median progression-free survival is the time to progression-free survival that corresponds to when the cumulative progression-free survival rate is 0.5, indicating that 50% of individuals will live through this time without disease progression.

SECONDARY OUTCOMES:
completion rate | Approximately 40 months from date of the first participant randomization
  The treatment completion rate is defined as the ratio of the number of patients actually completing the established intensity or number of cycles of treatment for subjects enrolled in the study to the total number of patients scheduled to complete the established intensity or number of cycles of treatment during the same period, in accordance with the conventional antineoplastic treatment schedule
Quality of Life(QoL) | Approximately 40 months from date of the first participant randomization
  Survival quality was compared by the Karnofsky Performance Status (KPS)score, a Karnofsky functional status rating scale.
median Overall Survival | Approximately 40 months from date of the first participant randomization
  Overall survival(OS) is defined as the period from the date of treatment to the date of death from any cause. The OS of patients who were alive at the last follow-up visit was counted as data censored at the time of the last follow-up visit. For patients who were lost to follow-up, their OS was data censored at the time of last confirmed survival prior to loss to follow-up. Median overall survival, which is the survival time corresponding to when the cumulative survival rate is 0.5, indicates that 50% of individuals will live beyond this time.
Disease Control Rate | Approximately 40 months from date of the first participant randomization
  Refers to the proportion of patients whose tumors shrink or are stable and remain so for a certain period of time, and includes cases of CR, PR and SD. Subjects had to be accompanied by a measurable tumor lesion at baseline, and the efficacy rating criteria were classified as complete remission (CR), partial remission (PR), stable disease (SD), and disease progression (PD) according to RECIST v1.1.
Objective Response Rate | Approximately 40 months from date of the first participant randomization
  Refers to the proportion of patients whose tumors have shrunk to a certain level and remained there for a certain period of time, and includes both CR and PR cases.
Duration of Response | Approximately 40 months from date of the first participant randomization
  Refers to the time from the first time the tumor was assessed as CR or PR (whichever was measured first) to the time of the first true recording of PD (using the smallest measurement recorded in the trial as a reference for disease progression).

CONTACTS AND LOCATIONS:
Locations (1):
- Renmin hosptial of Wuhan University, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Bray F, Ferlay J, Soerjomataram I, Siegel RL, Torre LA, Jemal A. Global cancer statistics 2018: GLOBOCAN estimates of incidence and mortality worldwide for 36 cancers in 185 countries. CA Cancer J Clin. 2018 Nov;68(6):394-424. doi: 10.3322/caac.21492. Epub 2018 Sep 12. PMID 30207593
- [Result] Chen W, Zheng R, Baade PD, Zhang S, Zeng H, Bray F, Jemal A, Yu XQ, He J. Cancer statistics in China, 2015. CA Cancer J Clin. 2016 Mar-Apr;66(2):115-32. doi: 10.3322/caac.21338. Epub 2016 Jan 25. PMID 26808342
- [Result] McCreery E, Costello J. Providing nutritional support for patients with cancer cachexia. Int J Palliat Nurs. 2013 Jan;19(1):32-7. doi: 10.12968/ijpn.2013.19.1.32. PMID 23354431
- [Result] Caillet P, Liuu E, Raynaud Simon A, Bonnefoy M, Guerin O, Berrut G, Lesourd B, Jeandel C, Ferry M, Rolland Y, Paillaud E. Association between cachexia, chemotherapy and outcomes in older cancer patients: A systematic review. Clin Nutr. 2017 Dec;36(6):1473-1482. doi: 10.1016/j.clnu.2016.12.003. Epub 2016 Dec 18. PMID 28017447
- [Result] Unsal D, Mentes B, Akmansu M, Uner A, Oguz M, Pak Y. Evaluation of nutritional status in cancer patients receiving radiotherapy: a prospective study. Am J Clin Oncol. 2006 Apr;29(2):183-8. doi: 10.1097/01.coc.0000198745.94757.ee. PMID 16601440
- [Result] Hill A, Kiss N, Hodgson B, Crowe TC, Walsh AD. Associations between nutritional status, weight loss, radiotherapy treatment toxicity and treatment outcomes in gastrointestinal cancer patients. Clin Nutr. 2011 Feb;30(1):92-8. doi: 10.1016/j.clnu.2010.07.015. Epub 2010 Aug 17. PMID 20719409
- [Result] Bourdeanu L, Frankel P, Yu W, Hendrix G, Pal S, Badr L, Somlo G, Luu T. Chemotherapy-induced nausea and vomiting in Asian women with breast cancer receiving anthracycline-based adjuvant chemotherapy. J Support Oncol. 2012 Jul-Aug;10(4):149-54. doi: 10.1016/j.suponc.2011.10.007. Epub 2012 Jan 4. PMID 22222249
- [Result] Serafini M, Jakszyn P, Lujan-Barroso L, Agudo A, Bas Bueno-de-Mesquita H, van Duijnhoven FJ, Jenab M, Navarro C, Palli D, Boeing H, Wallstrom P, Regner S, Numans ME, Carneiro F, Boutron-Ruault MC, Clavel-Chapelon F, Morois S, Grioni S, Panico S, Tumino R, Sacerdote C, Ramon Quiros J, Molina-Montes E, Huerta Castano JM, Barricarte A, Amiano P, Khaw KT, Wareham N, Allen NE, Key TJ, Jeurnink SM, Peeters PH, Bamia C, Valanou E, Trichopoulou A, Kaaks R, Lukanova A, Bergmann MM, Lindkvist B, Stenling R, Johansson I, Dahm CC, Overvad K, Jensen M, Olsen A, Tjonneland A, Lund E, Rinaldi S, Michaud D, Mouw T, Riboli E, Gonzalez CA. Dietary total antioxidant capacity and gastric cancer risk in the European prospective investigation into cancer and nutrition study. Int J Cancer. 2012 Aug 15;131(4):E544-54. doi: 10.1002/ijc.27347. Epub 2012 Jan 31. PMID 22072493
- [Result] Kolawole OM, Olatunji KT, Durowade KA. Molecular detection of human papillomavirus from abnormal cervical cytology of women attending a tertiary health facility in Ido-ekiti, southwest Nigeria. J Prev Med Hyg. 2016;57(2):E86-90. PMID 27582634
- [Result] Shitara K, Chin K, Yoshikawa T, Katai H, Terashima M, Ito S, Hirao M, Yoshida K, Oki E, Sasako M, Emi Y, Tsujinaka T. Phase II study of adjuvant chemotherapy of S-1 plus oxaliplatin for patients with stage III gastric cancer after D2 gastrectomy. Gastric Cancer. 2017 Jan;20(1):175-181. doi: 10.1007/s10120-015-0581-1. Epub 2015 Dec 1. PMID 26626800
- [Result] Climent M, Munarriz M, Blazeby JM, Dorcaratto D, Ramon JM, Carrera MJ, Fontane L, Grande L, Pera M. Weight loss and quality of life in patients surviving 2 years after gastric cancer resection. Eur J Surg Oncol. 2017 Jul;43(7):1337-1343. doi: 10.1016/j.ejso.2017.01.239. Epub 2017 Feb 9. PMID 28222970